CLINICAL TRIAL: NCT01771068
Title: Trial of a Parenting Discussion Group in Panama, Central America
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manchester (Other)
Collaborators: National Secretariat of Science, Technology and Innovation in Panama (SENACYT) (Unknown)
Responsible Party: Principal Investigator, Anilena Mejia, PhD Student, University of Manchester
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PTY12
Record Dates: First submitted 2013-01-11; First posted 2013-01-18 (Estimated); Last update posted 2013-01-18 (Estimated); Status verified 2013-01

CONDITIONS: Child Behavioural and Emotional Difficulties; Parenting Practices

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Waiting list (No Intervention)
- Parenting Discussion Group (Experimental): Two-hour discussion group on child noncompliance. Groups were composed by a maximum of 10 parents and were facilitated by the principal researcher, who is an accredited practitioner. The groups were interactive and discussion based, and a power point presentation with embedded-video clips was used to aid the facilitator. The key points covered in the discussion group included reasons for disobedience, parenting traps, encouraging good behaviour, and managing disobedience. Parents also received a workbook that included the content covered in the discussion group and 2 follow up telephone calls to check how they were doing after the discussion groups.
  Interventions: Behavioral: Triple P Positive Parenting Program Discussion Group "Dealing with Disobedience"

INTERVENTIONS:
Behavioral: Triple P Positive Parenting Program Discussion Group "Dealing with Disobedience"
  Arms: Parenting Discussion Group

SUMMARY:
The present study aims to examine the effectiveness of a parenting intervention, the Triple P Positive Parenting Program Level 3 discussion groups "dealing with disobedience". Triple P is a system of interventions to support families and was developed at the University of Queensland in Australia in the 1980's. As few studies have tested the effectiveness of parenting programs in developing countries, the present study took place in a developing country, Panama.

In a recent study carried out in Australia, this same intervention was found effective in reducing child behaviour problems and the use of dysfunctional parenting (Morawska, Haslam, Milne & Sanders, 2011).

DETAILED DESCRIPTION:
This is a randomized controlled trial (RCT) with two groups (waiting list versus Triple P discussion groups) and measurements at pre-intervention, post intervention, three and six months follow up.

The intervention trialed was a 2-hour, one-session discussion group on child noncompliance. Groups were composed by a maximum of 10 parents and were facilitated by the principal researcher, who is an accredited practitioner. The groups were interactive and discussion based, and a power point presentation with embedded-video clips were used to aid the facilitator. The key points that were covered in the discussion group included reasons for disobedience, parenting traps, encouraging good behaviour, and managing disobedience. Parents also received a workbook that included the content covered in the discussion group and 2 follow up telephone calls to check how they were doing after.

Participants were randomly assigned to a treatment group (Triple P discussion groups) or to a waiting list group. A statistician independent from the research team generated a random list of numbers. Randomization was stratified based on the level of child behavioural difficulties (high or low) measured at baseline. In order to ensure allocation concealment, sequentially-numbered, opaque, sealed envelopes (SNOSE) were opened after participants agreed to take part in the study and completed a baseline assessment. After randomization, those assigned to the waiting list group were assessed at time 1 (baseline) and then 4 weeks, 3 months and 6 months after the first assessment. Those assigned to the treatment group were assessed at time 1 (baseline), 2 weeks, 3 months and 6 months after the intervention. Assessments were carried out by a research assistant who was blind to group allocation.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be Panamanian
* must have at least one child between 3 and 12 years old
* must report some level of difficulty in dealing with their child behaviour.

Exclusion Criteria:

* no report of difficulty in dealing with child behaviour
* illiteracy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2012-04; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Change in Eyberg Child Behaviour Inventory (ECBI) | baseline, 2 weeks post intervention, 3 months and 6 months

SECONDARY OUTCOMES:
Change in Depression Anxiety Stress Scale 21 (DASS 21) | baseline, 2 weeks post intervention, 3 months and 6 months
Change in Parenting Scale (PS) | baseline, 2 weeks post intervention, 3 months and 6 months
Change in Parenting Task Checklist (PTC) | baseline, 2 weeks post intervention, 3 months and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Anilena Mejia, MSc, Principal Investigator — The University of Manchester; Rachel Calam, Professor, Principal Investigator — The University of Manchester; Matthew Sanders, Professor, Principal Investigator — The University of Queensland
Locations (1):
- Ministry of Education, District of Panama, Panama City, Provincia de Panamá, Panama